CLINICAL TRIAL: NCT00614952
Title: Diagnostic Validity Study and Cost Analysis of Domiciliary Respiratory
Brief Title: Cost/Effectiveness Analysis of the Respiratory Poligraphy at Home
Acronym: Telesleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PI 050444
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2012-12

CONDITIONS: Suspected Sleep Apnea; Daytime Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PR (Experimental)
  Interventions: Other: PR (respiratory polygraphy)
- PSG (Active Comparator)
  Interventions: Device: PSG (polysomnography)

INTERVENTIONS:
Device: PSG (polysomnography) — POLYSOMNOGRAPHY
  Arms: PSG
Other: PR (respiratory polygraphy) — respiratory polygraphy: level III of AASM
  Arms: PR

SUMMARY:
The abbreviated diagnostic sleep studies (RP), made at home and transferred telematically to the sleep laboratory, are useful for the diagnosis of sleep apnea and due to a lower cost, it could be an alternative to conventional polysomnography. Objectives: 1) Usefulness of domiciliary study evaluated by percentage of patients diagnosed of SAHS compared with PSG and agreement in the therapeutic decision. 2) Direct costs of patients included in the study. Design: controlled, randomized, crossed and blind (320 patients) comparing PR made at home with PSG, in patients suspicious of SAHS. The equipment transfer will be made by a transport agency from home to home in order to be universal the access to this diagnostic model. The file transmission with the raw data of the study will be made telematically by GPRS. If the aims of the study reach an end there will be a considerable change in the clinical practice making possible the international acceptation of domiciliary PR as diagnosis of SAHS and adapting the diagnosis of this syndrome to the new technologies of communication. The universalization of domiciliary PR would make possible that the diagnosis of SAHS could be done in any patient and in any country with GPRS technology and a transport agency, that is to say in all developed countries. As sleep apneas affect 5-7 million persons in Spain and there is association between sleep apneas and cardiovascular risk, in the immediate future we must evaluate this disease as we do today with the cholesterol determination. If our results are as predicted, the primary care physician could start and in a lot of cases finish the SAHS diagnostic process. This would simplify remarkably the diagnosis of SAHS and would alleviate a lot the process cost all over the world.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Without clinical suspicion referred to any other sleep pathology susceptible of presenting daytime sleepiness.
3. Living 20 Km or more far from the hospital participating in the study.

Exclusion Criteria:

1. Psychophysical incapacity to answer questionnaires.
2. Patients who do not get pass the proof of placing the PR (see below).
3. Patients who present restrictive chronic disease previously diagnosed (neoplasy, any origin chronic pain, renal failure, severe chronic obstructive pulmonary disease and any other limited chronic disease)
4. Structural cardiopaty or coronary documented non controlled by means of medical treatment .
5. Toxicomanies. Alcoholism (more than 80 gr/day in men and 60 gr/day in women.
6. Informed consent not obtained.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2006-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the two diagnostic models (PR at home and PSG) evaluated by means of percentage of patients who have established the diagnosis of SAHS and agreement in the therapeutic decision. | at the end of the study

SECONDARY OUTCOMES:
Direct and indirect cost of patients included in the study. | at the end of the study
Relationship cost/efficacy | at the end of study
Number of non valid studies in each group | at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Masa, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Hospital San Pedro de Alcántara. Servicio Extremeño de Salud, Cáceres, Caceres, Spain